CLINICAL TRIAL: NCT02211677
Title: Hemoglobin, Neutrophil to Lymphocyte Ratio and Platelet Count Improve Prognosis Prediction of TNM Staging System in Nasopharyngeal Carcinoma: A Prospective Multi-institutional Observation Study
Brief Title: Hemoglobin, Neutrophil to Lymphocyte Ratio and Platelet Count Improve Prognosis Prediction in Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yun-fei Xia, Department of Radiation Oncology, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Other Study IDs: B2014-002-01
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Nasopharyngeal Neoplasms; Blood Cell Count; Neoplasm Staging; Prognosis
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Low Risk Group: Each of the eight independent prognostic factors (age, sex, T and N stages, hemoglobin during radiotherapy, variation tendency of Hb, neutrophil-lymphocyte ratio before radiotherapy and platelet during radiotherapy) was assigned a number of points proportional to its regression coefficient to calculate prognostic index (PI), which ranged from 1 to 17. Patients with PI equal to 1-4 called the low risk group.
- Intermediate Risk Group: Each of the eight independent prognostic factors (age, sex, T and N stages, hemoglobin during radiotherapy, variation tendency of Hemoglobin, neutrophil-lymphocyte ratio before radiotherapy and platelet during radiotherapy) was assigned a number of points proportional to its regression coefficient to calculate prognostic index (PI), which ranged from 1 to 17. Patients with PI equal to 5-11 called the intermediate risk group.
- High Risk Group: Each of the eight independent prognostic factors (age, sex, T and N stages, hemoglobin during radiotherapy, variation tendency of Hemoglobin, neutrophil-lymphocyte ratio before radiotherapy and platelet during radiotherapy) was assigned a number of points proportional to its regression coefficient to calculate prognostic index (PI), which ranged from 1 to 17. Patients with PI equal to 12-17 called the high risk group.

SUMMARY:
RATIONALE

1. In patients with nasopharyngeal carcinoma, there is sometimes a discrepancy between actual clinical outcome and TNM stages because it is an anatomy-based system in which functional factors are not concerned.
2. Hemoglobin, neutrophil to lymphocyte ratio and platelet count were proved to improve prognosis prediction of TNM staging system in our previous retrospective study.

PURPOSE To validate that the prognostic index based on complete blood count and TNM system had higher prediction efficiency on survival in nasopharyngeal carcinoma than TNM system alone.

DETAILED DESCRIPTION:
Totally 720 patients with non-metastatic nasopharyngeal carcinoma will be include and will be divided into 3 groups (Low Risk, Intermediate Risk and High Risk Groups) according to their prognostic index, which is on basis of blood cell count indexes and TNM stage. The 3 groups of patients will undergo a radical radiotherapy or chemoradiotherapy and be followed until death or the end of the study. Comparison on survivals of the 3 groups will be made to validate the accuracy of the prognostic index. And comparison on prediction efficacy between prognostic index and TNM staging system will be made.

ELIGIBILITY:
Inclusion Criteria:

* Nasopharyngeal cancer patients diagnosed by pathology or cytology
* UICC/AJCC 2010 Stage T1-4 N0-3 M0
* Male or female patients with age between 18 and 75 years old
* Karnofsky Performance Scores ≥ 60
* Expected survival ≥ 3 months
* Without dysfunction of heart, lung, liver, kidney and hematopoiesis

Exclusion Criteria:

* Karnofsky Performance Status Score < 70'
* Radiotherapy uncompleted (≥ 1 fraction missing)
* Distant metastases before or during radiotherapy
* Without weekly complete blood count during radiotherapy
* Application of colony stimulating factor such as erythropoietin
* Signs of infection before radiotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the participants involved in our study are patients who are first diagnosed nasopharyngeal carcinoma pathologically and treated with radical radiotherapy or chemoradiotherapy in ourhospital from August 1st 2014 to July 31st 2015.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 years after diagnosis
  The period until any event (death, local recurrence or distant metastasis) is detected.

SECONDARY OUTCOMES:
5-year disease-free survival | 5 years after diagnosis
  The period until local recurrence or distant metastasis is detected.
5-year recurrence-free survival | 5 years after diagnosis
  The period until local recurrence is detected.
5-year distant-free survival | 5 years after diagnosis
  The period until distant metastasis is detected.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, MD, Principal Investigator — Sun Yat-sen University
Locations (6):
- China (6):
  - The Fisrt Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Province Hospital, Hefei, Anhui
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Central Hospital of Shaoyang, Shaoyang, Hunan
  - The Affiliated Hospital of Luzhou Medical College, Luzhou, Sichuan